CLINICAL TRIAL: NCT02872311
Title: Open-Label, Randomized Study of Immune Response to Licensed Influenza Vaccines in Adults 65-74 Years of Age (US Flu Vaccine Effectiveness Serologic Study, 2016-17 and 2017-18)
Brief Title: Open-Label Influenza Vaccine Evaluation
Acronym: OLIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marshfield Clinic Research Foundation (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Huong Nguyen, PhD, Research Scientist, Marshfield Clinic Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MCL10416
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Results first posted 2019-12-19 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Immune Response
Keywords: Vaccine; Influenza; High Dose; Adjuvanted; Recombinant
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluBlok

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- High Dose Influenza Vaccine (Active Comparator): This group will be administered High Dose (HD) influenza vaccination (0.5 mL intramuscular (IM) injection) in the first and second years of the study.
  Interventions: Biological: High Dose Influenza vaccine
- Adjuvanted Influenza Vaccine (Active Comparator): This group will be administered adjuvanted influenza vaccination (0.5 mL intramuscular (IM) injection) in the first and second years of the study.
  Interventions: Biological: Adjuvanted Influenza vaccine
- Standard Dose Influenza Vaccine+HD (Active Comparator): This group will be administered standard dose flu vaccination (0.5 mL intramuscular (IM) injection) in the first year of the study and high dose influenza vaccine (0.5 mL intramuscular (IM) injection) in the second year of the study.
  Interventions: Biological: High Dose Influenza vaccine; Biological: Standard Dose Influenza vaccine
- Standard Dose Influenza Vaccine +Adj (Active Comparator): This group will be administered standard dose flu vaccination (0.5 mL intramuscular (IM) injection) in the first year and adjuvanted influenza vaccination (0.5 mL intramuscular (IM) injection) in the second year of the study.
  Interventions: Biological: Adjuvanted Influenza vaccine; Biological: Standard Dose Influenza vaccine
- Standard Dose Influenza Vaccine+Recomb (Active Comparator): This group will be administered a standard dose flu vaccination (0.5 mL intramuscular (IM) injection) in the first year and recombinant influenza vaccination (0.5 mL intramuscular (IM) injection) in the second year of the study.
  Interventions: Biological: Standard Dose Influenza vaccine; Biological: Recombinant Influenza vaccine

INTERVENTIONS:
Biological: High Dose Influenza vaccine — Licensed and FDA approved Fluzone HD vaccine to be administered to study participants
  Other Names: Fluzone HD
  Arms: High Dose Influenza Vaccine; Standard Dose Influenza Vaccine+HD
Biological: Adjuvanted Influenza vaccine — Licensed and FDA approved FluAd vaccine to be administered to study participants
  Other Names: FluAd
  Arms: Adjuvanted Influenza Vaccine; Standard Dose Influenza Vaccine +Adj
Biological: Standard Dose Influenza vaccine — Licensed and FDA approved Fluvirin vaccine to be administered to study participants
  Other Names: Fluvirin Standard Dose
  Arms: Standard Dose Influenza Vaccine +Adj; Standard Dose Influenza Vaccine+HD; Standard Dose Influenza Vaccine+Recomb
Biological: Recombinant Influenza vaccine — Licensed and FDA approved FluBlok vaccine to be administered to study participants
  Other Names: FluBlok
  Arms: Standard Dose Influenza Vaccine+Recomb

SUMMARY:
This is an open-label, randomized trial in up to 210 adults aged 65-74 years to evaluate the immune response to consecutive influenza vaccination across 2 seasons. Participants will be randomized to receive 1 of 3 licensed and recommended vaccines in the first year; 2 arms will receive the same vaccination in the second year and the third arm will be randomized again to 1 of 3 licensed vaccines. All participants will have pre and post-vaccination serum blood draws for a total of 6 draws over 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-74 years at the time of study enrollment and are ambulatory and live in selected Wisconsin community or surrounding communities.
* Willing and able to give informed consent prior to study enrollment
* Able to comply with study requirements.

Exclusion Criteria:

* Prior receipt of 2016-17 influenza vaccine
* Current participation in another clinical trial
* Presence of a contraindication to influenza vaccine

Ages: 65 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 179 (Actual)
Dates: Start 2016-09; Primary Completion 2018-04 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McLean HQ, Levine MZ, King JP, Flannery B, Belongia EA. Serologic response to sequential vaccination with enhanced influenza vaccines: Open label randomized trial among adults aged 65-74 years. Vaccine. 2021 Dec 3;39(49):7146-7152. doi: 10.1016/j.vaccine.2021.10.072. Epub 2021 Nov 10. PMID 34774360

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard+High Dose: This group will be administered standard influenza vaccination (0.5 mL intramuscular (IM) injection) in the first year and high dose influenza vaccination (0.5mL intramuscular (IM) injection) in the second year of the study.
  Standard Dose Influenza vaccine: Licensed and FDA approved Fluvirin vaccine to be administered to study participants.
  High Dose Influenza vaccine: Licensed and FDA approved Fluzone HD vaccine to be administered to study participants
- Standard+Adjuvanted: This group will be administered standard influenza vaccination (0.5 mL intramuscular (IM) injection) in the first year and adjuvanted influenza vaccination (0.5 mL intramuscular (IM) injection) in the second year of the study.
  Standard Dose Influenza vaccine: Licensed and FDA approved Fluvirin vaccine to be administered to study participants.
  Adjuvanted Influenza vaccine: Licensed and FDA approved FluAd vaccine to be administered to study participants
- Standard+Recombinant: This group will be administered standard influenza vaccination (0.5 mL intramuscular (IM) injection) in the first year and recombinant influenza vaccination (0.5 mL intramuscular (IM) injection) in the second year of the study.
  Standard Dose Influenza vaccine: Licensed and FDA approved Fluvirin vaccine to be administered to study participants.
  Recombinant Influenza vaccine: Licensed and FDA approved FluBlok vaccine to be administered to study participants
Period: Overall Study
Arm/Group | High Dose Influenza Vaccine | Adjuvanted Influenza Vaccine | Standard+High Dose | Standard+Adjuvanted | Standard+Recombinant
Started | 59 | 60 | 20 | 20 | 20
Completed | 55 | 58 | 19 | 20 | 20
Not Completed | 4 | 2 | 1 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Influenza Vaccine | Adjuvanted Influenza Vaccine | Standard Dose Influenza Vaccine+HD | Standard Dose Influenza Vaccine +Adj | Standard Dose Influenza Vaccine+Recomb | Total
Number analyzed (Participants) | 55 | 58 | 19 | 20 | 20 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (2.7) | 69.6 (2.6) | 69.4 (2.9) | 69.2 (2.2) | 70 (2.7) | 70 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 33 | 10 | 12 | 9 | 90
  Male | 29 | 25 | 9 | 8 | 11 | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race : White | 55 | 58 | 19 | 20 | 20 | 172
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55 | 58 | 19 | 20 | 20 | 172

OUTCOME MEASURES:

1. Primary Outcome: HI Titers, HD vs. AD, Yr 1 Day 28 Post Vaccination
Description: Hemagglutination Inhibition (HI) titers to vaccine viruses for high dose and adjuvanted vaccine recipients at 28 days post vaccination 2016-17
Time Frame: Year 1, Day 28 post vaccination
Population: This primary objective evaluated only recipients in the arms receiving high dose and adjuvanted vaccine in year 1.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | High Dose Influenza Vaccine | Adjuvanted Influenza Vaccine
Number analyzed (Participants) | 55 | 58
Titer
  A/H1/California | 175 [128 to 239] | 117 [87 to 159]
  A/H3/Hong Kong | 144 [102 to 201] | 118 [87 to 159]
  B/Brisbane(Victoria) | 166 [117 to 236] | 81 [59 to 112]

2. Primary Outcome: HI Titers, HD vs. AD, Yr 1 Day 182 Post Vaccination
Description: Hemagglutination Inhibition (HI) titers to vaccine viruses for high dose and adjuvanted vaccine recipients at 182 days post vaccination 2016-17
Time Frame: Year 1, Day 182 post vaccination
Population: This primary objective evaluated only recipients in the arms receiving high dose and adjuvanted vaccine in year 1.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | High Dose Influenza Vaccine | Adjuvanted Influenza Vaccine
Number analyzed (Participants) | 55 | 58
Titer
  A/H1/California | 83 [62 to 110] | 56 [41 to 77]
  A/H3/Hong Kong | 83 [60 to 113] | 68 [51 to 91]
  B/Brisbane(Victoria) | 61 [43 to 88] | 44 [33 to 60]

3. Primary Outcome: HI Titers, HD vs. AD, Yr 1 Day 365 Post Vaccination
Description: Hemagglutination Inhibition (HI) titers to vaccine viruses for high dose and adjuvanted vaccine recipients at 365 days post vaccination 2016-17
Time Frame: Year 1, Day 365 post vaccination
Population: This primary objective evaluated only recipients in the arms receiving high dose and adjuvanted vaccine in year 1.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | High Dose Influenza Vaccine | Adjuvanted Influenza Vaccine
Number analyzed (Participants) | 55 | 58
Titer
  A/H1/California | 54 [40 to 72] | 44 [32 to 60]
  A/H3/Hong Kong | 75 [55 to 103] | 75 [57 to 100]
  B/Brisbane(Victoria) | 36 [25 to 52] | 24 [17 to 32]

4. Primary Outcome: HI Titers, HD vs. AD, Yr 2 Day 28 Post Vaccination
Description: Hemagglutination Inhibition (HI) titers to vaccine viruses for high dose and adjuvanted vaccine recipients at 28 days post vaccination 2017-18
Time Frame: Year 2, Day 28 post vaccination
Population: This primary objective evaluated only recipients in the arms receiving high dose and adjuvanted vaccine in year 1.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | High Dose Influenza Vaccine | Adjuvanted Influenza Vaccine
Number analyzed (Participants) | 55 | 58
Titer
  A/H1/Michigan | 83 [64 to 107] | 101 [74 to 139]
  A/H3/Hong Kong | 158 [114 to 220] | 158 [123 to 203]
  B/Brisbane(Victoria) | 63 [46 to 87] | 45 [33 to 61]

5. Primary Outcome: HI Titers, HD vs. AD, Yr 2 Day 182 Post Vaccination
Description: Hemagglutination Inhibition (HI) titers to vaccine viruses for high dose and adjuvanted vaccine recipients at 182 days post vaccination 2017-18
Time Frame: Year 2, Day 182 post vaccination
Population: This primary objective evaluated only recipients in the arms receiving high dose and adjuvanted vaccine in year 1.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | High Dose Influenza Vaccine | Adjuvanted Influenza Vaccine
Number analyzed (Participants) | 55 | 58
Titer
  A/H1/Michigan | 46 [35 to 61] | 44 [32 to 61]
  A/H3/Hong Kong | 101 [74 to 138] | 124 [93 to 165]
  B/Brisbane(Victoria) | 44 [31 to 61] | 30 [22 to 42]

6. Secondary Outcome: HI Response by Prior Season Vaccination, Yr 1, Day 28 Post Vaccination
Description: Hemagglutination inhibition (HI) Titers by prior season (2015-16) vaccination status among adjuvant and high dose vaccine recipients 28 days post vaccination, 2016-17
Time Frame: Year 1, Day 28 post vaccination
Population: Secondary objective examines response in adjuvant and high dose recipients by prior season vaccination status.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- IIV-ADJ: 2015-16 Standard dose vaccine recipient who received adjuvanted vaccine in the study in 2016-17
- IIV-HD: 2015-16 Standard dose vaccine recipient who received high dose vaccine in the study in 2016-17
- None-ADJ: 2015-16 Unvaccinated individual who received adjuvanted vaccine in the study in 2016-17
- None-HD: 2015-16 Unvaccinated individual who received high dose vaccine in the study in 2016-17
Arm/Group | IIV-ADJ | IIV-HD | None-ADJ | None-HD
Number analyzed (Participants) | 44 | 40 | 14 | 15
Titer
  A/H1/California | 116 [82 to 165] | 136 [95 to 193] | 122 [62 to 241] | 343 [194 to 608]
  A/H3/Hong Kong | 105 [76 to 147] | 128 [85 to 193] | 168 [82 to 343] | 197 [106 to 366]
  B/Brisbane(Victoria) | 62 [45 to 84] | 142 [93 to 217] | 195 [87 to 435] | 254 [136 to 475]

7. Secondary Outcome: HI Response by Prior Season Vaccination, Yr 1, Day 182 Post Vaccination
Description: Hemagglutination inhibition (HI) Titers by prior season (2015-16) vaccination status among adjuvant and high dose vaccine recipients 182 days post vaccination, 2016-17
Time Frame: Year 1, Day 182 post vaccination
Population: Secondary objective examines response in adjuvant and high dose recipients by prior season vaccination status.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | IIV-ADJ | IIV-HD | None-ADJ | None-HD
Number analyzed (Participants) | 44 | 40 | 14 | 15
Titer
  A/H1/California | 59 [41 to 85] | 67 [49 to 91] | 48 [23 to 98] | 146 [81 to 264]
  A/H3/Hong Kong | 68 [49 to 96] | 84 [56 to 126] | 67 [35 to 128] | 78 [47 to 129]
  B/Brisbane(Victoria) | 36 [27 to 48] | 51 [33 to 77] | 86 [38 to 196] | 103 [52 to 202]

8. Secondary Outcome: HI Response by Prior Season Vaccination, Yr 1, Day 365 Post Vaccination
Description: Hemagglutination inhibition (HI) Titers by prior season (2015-16) vaccination status among adjuvant and high dose vaccine recipients 365 days post vaccination, 2016-17
Time Frame: Year 1, Day 365 post vaccination
Population: Secondary objective examines response in adjuvant and high dose recipients by prior season vaccination status.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | IIV-ADJ | IIV-HD | None-ADJ | None-HD
Number analyzed (Participants) | 44 | 40 | 14 | 15
Titer
  A/H1/California | 51 [36 to 74] | 48 [34 to 67] | 26 [13 to 52] | 73 [39 to 137]
  A/H3/Hong Kong | 82 [59 to 114] | 79 [53 to 117] | 58 [31 to 107] | 66 [38 to 117]
  B/Brisbane(Victoria) | 20 [15 to 28] | 34 [22 to 52] | 38 [17 to 86] | 44 [20 to 96]

9. Secondary Outcome: MN Titers, HD vs. AD, Year 1, Day 28 Post Vaccination
Description: Microneutralization antibody titers to vaccine and drifted viruses among high dose and adjuvanted vaccine recipients 28 days post vaccination, 2016-17
Time Frame: Year 1, Day 28 post vaccination
Population: Secondary objective examines response in adjuvant and high dose recipients to vaccine and drifted viruses.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | High Dose Influenza Vaccine | Adjuvanted Influenza Vaccine
Number analyzed (Participants) | 55 | 58
Titer
  A/H3/Hong Kong 4801 (egg) | 256 [175 to 373] | 246 [160 to 380]
  A/H3/Hong Kong 4801 (siat cell) | 57 [42 to 79] | 69 [49 to 96]
  A/H3/NZ0783 (siat cell) | 47 [33 to 66] | 52 [37 to 71]
  A/H3/OR19 (siat cell) | 32 [22 to 46] | 39 [27 to 56]

10. Secondary Outcome: MN Titers, HD vs. AD, Year 1, Day 182 Post Vaccination
Description: Microneutralization antibody titers to vaccine and drifted viruses among high dose and adjuvanted vaccine recipients 182 days post vaccination, 2016-17
Time Frame: Year 1, Day 182 post vaccination
Population: Secondary objective examines response in adjuvant and high dose recipients to vaccine and drifted viruses.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | High Dose Influenza Vaccine | Adjuvanted Influenza Vaccine
Number analyzed (Participants) | 55 | 58
Titer
  A/H3/Hong Kong 4801 (egg) | 138 [91 to 208] | 132 [89 to 196]
  A/H3/Hong Kong 4801 (siat cell) | 44 [33 to 60] | 42 [30 to 59]
  A/H3/NZ0783 (siat cell) | 29 [22 to 40] | 30 [22 to 41]
  A/H3/OR19 (siat cell) | 24 [18 to 33] | 25 [18 to 36]

11. Secondary Outcome: MN Titers, HD vs. AD, Year 1, Day 365 Post Vaccination
Description: Microneutralization antibody titers to vaccine and drifted viruses among high dose and adjuvanted vaccine recipients 365 days post vaccination, 2016-17
Time Frame: Year 1, Day 365 post vaccination
Population: Secondary objective examines response in adjuvant and high dose recipients to vaccine and drifted viruses.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | High Dose Influenza Vaccine | Adjuvanted Influenza Vaccine
Number analyzed (Participants) | 55 | 58
Titer
  A/H3/Hong Kong 4801 (egg) | 138 [91 to 207] | 132 [89 to 196]
  A/H3/Hong Kong 4801 (siat cell) | 45 [33 to 60] | 55 [51 to 74]
  A/H3/NZ0783 (siat cell) | 29 [22 to 40] | 30 [22 to 41]
  A/H3/OR19 (siat cell) | 24 [18 to 33] | 25 [18 to 36]

12. Secondary Outcome: MN Titers (A/Hong Kong (Siat Cell)), HD vs. AD, Year 2, Day 28 Post Vaccination
Description: Microneutralization antibody titers to vaccine virus (A/Hong Kong (siat cell) among high dose and adjuvanted vaccine recipients 28 days post vaccination, 2017-18
Time Frame: Year 2, Day 28 post vaccination
Population: Secondary objective examines response in adjuvant and high dose recipients to A/Hong Kong (siat cell) virus in year 2, post vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | High Dose Influenza Vaccine | Adjuvanted Influenza Vaccine
Number analyzed (Participants) | 55 | 58
Titer | 73 [55 to 96] | 95 [71 to 125]

13. Secondary Outcome: HI Titers, HD vs. AD vs. RIV With Prior Season Standard (IIV) Dose, Year 2, Day 28 Post Vaccination
Description: Hemagglutination Inhibition (HI) titers to vaccine viruses among adjuvant, high dose and recombinant recipients with prior season standard dose vaccine at 28 days post vaccination 2017-18
Time Frame: Year 2, Day 28 post vaccination
Population: This secondary objective aimed to look at subjects receiving standard dose vaccine in the previous season and one of 3 licensed vaccines in the 2017-18 season.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Standard Dose Influenza Vaccine +Adj | Standard Dose Influenza Vaccine+HD | Standard Dose Influenza Vaccine+Recomb
Number analyzed (Participants) | 20 | 19 | 20
Titer
  A/H1/Michigan | 44 [24 to 81] | 86 [48 to 154] | 126 [68 to 232]
  A/H3/Hong Kong | 126 [72 to 220] | 163 [84 to 317] | 174 [97 to 313]
  B/Brisbane(Victoria) | 35 [21 to 57] | 83 [42 to 164] | 53 [30 to 94]

14. Secondary Outcome: HI Titers, HD vs. AD vs. RIV With Prior Season Standard (IIV) Dose, Year 2, Day 182 Post Vaccination
Description: Hemagglutination Inhibition (HI) titers to vaccine viruses among adjuvant, high dose and recombinant recipients with prior season standard dose vaccine at 182 days post vaccination 2017-18
Time Frame: Year 2, Day 182 post vaccination
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Standard Dose Influenza Vaccine +Adj | Standard Dose Influenza Vaccine+HD | Standard Dose Influenza Vaccine+Recomb
Number analyzed (Participants) | 20 | 19 | 20
Titer
  A/H1/Michigan | 26 [15 to 45] | 33 [17 to 66] | 75 [41 to 135]
  A/H3/Hong Kong | 95 [55 to 164] | 122 [67 to 222] | 135 [75 to 242]
  B/Brisbane(Victoria) | 26 [16 to 41] | 47 [26 to 86] | 33 [19 to 58]

15. Secondary Outcome: HI Titers, IIV+AD or HD vs. Sequential AD or HD, Year 2, Day 28 Post Vaccination
Description: Hemagglutination inhibition (HI) titers among HD and AD based on prior season vaccination (standard or sequential same vaccination) at 28 days after vaccination, 2017-18
Time Frame: Year 2, Day 28 post vaccination
Population: This secondary objective selects individuals receiving high dose or adjuvanted vaccine in year 2 of the study and compares immune response by vaccine received in the prior season.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Adjuvant Influenza Vaccine: This group will be administered adjuvanted influenza vaccination (0.5 mL intramuscular (IM) injection) in the first and second years of the study.
  Adjuvanted Influenza vaccine: Licensed and FDA approved FluAd vaccine to be administered to study participants
Arm/Group | Adjuvant Influenza Vaccine | High Dose Influenza Vaccine | Standard Dose Influenza Vaccine +Adj | Standard Dose Influenza Vaccine+HD
Number analyzed (Participants) | 58 | 55 | 20 | 19
Titer
  A/H1/Michigan | 101 [74 to 139] | 83 [64 to 107] | 44 [24 to 81] | 86 [48 to 154]
  A/H3/Hong Kong | 158 [123 to 203] | 158 [114 to 220] | 126 [72 to 220] | 163 [84 to 317]
  B/Brisbane(Victoria) | 45 [33 to 61] | 63 [46 to 87] | 35 [21 to 57] | 83 [42 to 164]

16. Secondary Outcome: HI Titers, IIV+AD or HD vs. Sequential AD or HD, Year 2, Day 182 Post Vaccination
Description: Hemagglutination inhibition (HI) titers among HD and AD based on prior season vaccination (standard or sequential same vaccination) at 182 days after vaccination, 2017-18
Time Frame: Year 2, Day 182 post vaccination
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Adjuvant Influenza Vaccine | High Dose Influenza Vaccine | Standard Dose Influenza Vaccine +Adj | Standard Dose Influenza Vaccine+HD
Number analyzed (Participants) | 58 | 55 | 20 | 19
Titer
  A/H1/Michigan | 44 [32 to 61] | 46 [35 to 51] | 26 [15 to 45] | 33 [17 to 66]
  A/H3/Hong Kong | 124 [93 to 165] | 101 [74 to 138] | 95 [55 to 164] | 122 [67 to 222]
  B/Brisbane(Victoria) | 30 [22 to 42] | 44 [31 to 61] | 26 [16 to 41] | 47 [26 to 86]

17. Secondary Outcome: Number of Participants With Vaccine Failure, Year 1
Description: Number of Participants with Vaccine Failure in Year 1 by vaccine type
Time Frame: Year 1, Post season
Population: Results of influenza surveillance after the first year examines individuals by the vaccine type received in Year 1.
Measure: Count of Participants; unit: Participants
Groups:
- High Dose Influenza Vaccine: This group received High Dose vaccine in the first year of the study.
- Adjuvanted Influenza Vaccine: This group received adjuvanted vaccine in the first year of the study.
- Standard Dose Influenza Vaccine: This group received standard dose in the first year of the study.
Arm/Group | High Dose Influenza Vaccine | Adjuvanted Influenza Vaccine | Standard Dose Influenza Vaccine
Number analyzed (Participants) | 55 | 58 | 59
Participants
  H3 Positive | 4 | 3 | 1
  B Positive | 0 | 1 | 1

18. Secondary Outcome: Number of Participants With Vaccine Failure, Year 2
Description: Number of Participants with Vaccine Failure in Year 2 by two-year vaccine history
Time Frame: Year 2, Post season
Population: Results of influenza surveillance after the second year examines individuals by groups based on the vaccine types received in both seasons.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Influenza Vaccine | Adjuvanted Influenza Vaccine | Standard+High Dose | Standard+Adjuvanted | Standard+Recombinant
Number analyzed (Participants) | 55 | 58 | 19 | 20 | 20
Participants
  H3 positive | 3 | 6 | 1 | 2 | 3
  B positive | 4 | 1 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: 18 months of the study
Arm/Group | High Dose Influenza Vaccine | Adjuvanted Influenza Vaccine | Standard Dose Influenza Vaccine+HD | Standard Dose Influenza Vaccine +Adj | Standard Dose Influenza Vaccine+Recomb
All-Cause Mortality (participants affected / at risk) | 2/55 | 0/58 | 0/19 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/58 | 0/19 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/55 | 0/58 | 0/19 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT02872311/Prot_SAP_000.pdf